CLINICAL TRIAL: NCT01893567
Title: Subject Reported Target-lesion Numeric Rating Scale Evaluation by Subjects With Plaque Psoriasis Treated With Clobex® (Clobetasol Propionate) Spray 0.05%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLI.04.SPR.US10243
Record Dates: First submitted 2013-06-26; First posted 2013-07-09 (Estimated); Results first posted 2014-07-11 (Estimated); Last update posted 2022-09-27 (Actual); Status verified 2018-08

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Clobex spray (Experimental)
  Interventions: Drug: Clobex Spray

INTERVENTIONS:
Drug: Clobex Spray
  Other Names: Clobetasol propionate spray

SUMMARY:
The aim of this study is to investigate the utility of a technological based rating scale for assessing improvement in plaque psoriasis with Clobex spray treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older.
* Subjects with a board certified dermatologist clinical diagnosis of active moderate to severe psoriasis lesions affecting up to 20% of the body surface area at the baseline visit, and in the opinion of the investigator, is otherwise a good candidate for treatment with clobetasol propionate 0.05% spray.
* Subjects with a target lesion of at least 1 cm x 1 cm
* Subjects who agree to be photographed at each visit

Exclusion Criteria:

* Subjects with any condition or presentation that may, in the opinion of the investigator, may put the subject at risk, may confound study results, or may interfere with participation in the study.
* Subjects with any known allergies to any of the ingredients listed on the test article label or surgical ink.
* Subjects who are pregnant or breast-feeding, or who plan to become pregnant or breast feed during the course of the trial.
* Subjects that are relatives of the investigator, or are themselves or a relative of any study staff or any Galderma employee.
* Subjects who have participated in an investigational study within 30 days of enrollment; participated in biologic investigational studies within 90 days of enrollment, or subjects planning to participate in any other interventional clinical research study while enrolled in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fasahat Hamzavi, MD, Principal Investigator — Hamzavi Dermatology
Locations (1):
- Hamzavi Dermatology, Fort Gratiot, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Clobex Spray: Clobex Spray
Period: Overall Study
Arm/Group | Clobex Spray
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Clobex Spray
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Subject Reported Target Lesion Severity Score.
Description: Subject reported mean scores of the target lesion numeric rating scale (TL-NRS; scale of 0 (no psoriasis) to 10 (very severe psoriasis)) at end of study.
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clobex Spray
Number analyzed (Participants) | 28
units on a scale | 4.0 (2.5)

2. Secondary Outcome: Investigator Reported Target Lesion Severity Score
Description: Investigator reported mean scores of the target lesion numeric rating scale (TL-NRS; scale of 0 (no psoriasis) to 10 (very severe psoriasis)) at end of study
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Clobex Spray
Number analyzed (Participants) | 28
units on a scale | 3.3 (2.1)

ADVERSE EVENTS:
Time Frame: From baseline up to Day 15
Arm/Group | Clobex Spray
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 4/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobex Spray (N=28)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin plaque (Skin and subcutaneous tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No